CLINICAL TRIAL: NCT00243022
Title: Phase II Randomized Evaluation of 5-Lipoxygenase Inhibition by Herbal Complementary and Alternative Medicine Approach Compared to Control as an Adjuvant Therapy in Newly Diagnosed and Recurrent High-grade Gliomas
Brief Title: Dietary, Herbal and Alternative Medicine in Glioblastoma Multiforme
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Ali Altunkaya (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Ali Altunkaya, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE1304; CCF-7348 (Other: Cleveland Clinic IRB); NCI-2010-01384 (Other: NCI/CTRP); R21CA107277-01 (NIH)
Record Dates: First submitted 2005-10-20; First posted 2005-10-21 (Estimated); Results first posted 2013-07-30 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Brain and Central Nervous System Tumors; Cerebral Edema
Keywords: cerebral edema; adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Edema; Glioblastoma; Gliosarcoma; Astrocytoma; Oligodendroglioma | interventions — Frankincense; Vitamin B 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (intervention) (Experimental): Patients receive oral Boswellia serrata extract 4 times a day and oral cyanocobalamin (vitamin B 12) once a day for 6 months in the absence of unacceptable toxicity.
  Interventions: Drug: Boswellia serrata extract; Dietary Supplement: cyanocobalamin
- Arm II (control) (Active Comparator): Patients in the control arm receive oral cyanocobalamin (vitamin B 12) once a day for 6 months.
  Interventions: Dietary Supplement: cyanocobalamin

INTERVENTIONS:
Drug: Boswellia serrata extract — given orally
  Arms: Arm I (intervention)
Dietary Supplement: cyanocobalamin — given orally
  Other Names: Vitamin B12

SUMMARY:
RATIONALE: Giving the herb Boswellia serrata after surgery and radiation therapy may slow the growth of any remaining tumor cells. It is not yet known whether giving Boswellia serrata together with standard treatment is more effective than standard treatment alone in treating high-grade gliomas.

PURPOSE: This randomized phase II trial is the study of a combination of complementary and alternative medicine (CAM) herbal supplement intervention as an adjuvant to standard treatment of patients with newly diagnosed and recurrent high-grade gliomas (HGG). The central hypothesis of this application is that a herbal preparation that inhibits 5-LO activity, will produce measurable biologically meaningful decrease in 5-LO eicosanoid production and brain edema that will be associated with improved survival and quality of life in patients with HGG.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether a herbal approach to decreasing 5-LO eicosanoid production reduces peritumoral brain edema in patients with HGG.

Secondary

* To determine if this adjuvant approach improves the quality of life and progression free and overall survival of patients with HGG.

OUTLINE: This a randomized, controlled study. Patients are randomized to 1 of 2 treatment arms.

* Arm I (intervention): Patients receive oral Boswellia serrata herbal extract 4 times a day and oral cyanocobalamin (vitamin B-12) once a day for 6 months in the absence of unacceptable toxicity.
* Arm II (control): Patients receive oral vitamin B-12 once a day for 6 months. All patients are encouraged to eat a regular balanced diet (as recommended by the American Cancer Society for cancer prevention) with limited consumption of red and processed meats.

Quality of life will be assessed at baseline and then at 2, 4, 6, 12, and 24 months.

After completion of study treatment, patients will be followed every 6 months.

PROJECTED ACCRUAL: A total of 70 patients (35 per treatment arm) will be accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients after surgical removal of histologically confirmed World Health Organization high-grade gliomas, including astrocytomas grade III (anaplastic astrocytoma), astrocytoma grade IV (glioblastoma multiforme, GBM), anaplastic oligodendroglioma and oligoastrocytoma
* Karnofsky performance status of greater or equal 60
* Patients who signed informed consent
* Patients can be receiving standard or investigational chemotherapy , hormonal therapy, immunotherapy or biologic agents as the primary treatment for their tumor
* Glucocorticoid therapy is allowed
* Bone marrow function (absolute neutrophil count [ANC] >=1500/mm^3 and platelet count >=75,000/mm^3); in the event of plate count dropping below 50,000/ mm^3 the Boswellia will be withdrawn until plate count reaches 75,000 mm^3 and above
* Liver function (bilirubin and alkaline phosphatase =< 2 x normal and serum glutamic oxaloacetic transaminase [SGOT] =< 3 x normal)
* Renal function (blood urea nitrogen [BUN] or creatinine =< 1.5 x normal)
* Patients suffering from mild to moderate asthma, liver and kidney disease; an assessment of the condition will be made to establish a baseline and monitor progress at 4 weekly intervals to start with for the first two months and thereafter at the usual study intervals of 4 and 6 months; if there is any significant deterioration in their condition the Boswellia will be withdrawn until these parameters are restored to their pre-treatment levels

EXCLUSION CRITERIA:

* Any medical condition that could interfere with eating and oral administration of B. serrata
* Patients already taking herbal preparations that contain 5-LO inhibitors
* Any previous (within the past 3 years) or concurrent malignancies at other sites, with the exception of surgically cured carcinoma-in-situ of the cervix and non-melanoma skin cancer
* Pregnancy and breastfeeding
* Active infection
* Inability to be followed closely at the Cleveland Clinic Foundation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-09; Primary Completion 2010-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glen Stevens, DO, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from September 2004-September 2010 from local medical clinic.
Groups:
- Arm I (Intervention): Patients receive oral Boswellia serrata extract 4 times a day and oral cyanocobalamin (vitamin B 12) once a day for 6 months in the absence of unacceptable toxicity.
  cyanocobalamin : 50 ug/day given orally
  Boswellia serrata extract : 4x (3-12.5) ml/day given orally, that is 720-3000mg of total Boswellic acids (three isomers)/day
- Arm II (Control): Patients in the control arm receive oral cyanocobalamin (vitamin B 12) once a day for 6 months.
  cyanocobalamin : 50 ug/day given orally
Period: Overall Study
Arm/Group | Arm I (Intervention) | Arm II (Control)
Started | 7 | 5
Completed | 5 | 4
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 1 | 0
Not completed — Difficult Travel Distance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm II (Control): Patients in the control arm receive oral cyanocobalamin (vitamin B 12) once a day for 6 months.
  cyanocobalamin : 50 ug/daygiven orally
- Total: Total of all reporting groups
Arm/Group | Arm I (Intervention) | Arm II (Control) | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Customized [Number; unit: participants]
  30-39 years | 1 | 0 | 1
  40-49 years | 3 | 3 | 6
  50-59 years | 1 | 2 | 3
  60-69 years | 1 | 0 | 1
  70-79 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 5 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 4 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 5 | 12
Baseline edema measure [Mean (Standard Deviation); unit: cm^3] — Baseline measure was acquired for 11 patients. Six on Arm I and five on Arm II.
  cm^3 | 10.8 (11.1) | 11.3 (8.1) | 11.1 (9.4)

OUTCOME MEASURES:

1. Primary Outcome: Change From Pooled Baseline in Peritumoral Brain Edema
Description: The relative change from baseline will be assessed longitudinally, however, the main comparison of interest is the relative change at the 4-month evaluation. For each patient change = edema at follow up - baseline edema
Time Frame: at 2 months
Population: Patients with baseline and follow up peritumoral edema measurement. Closest measurement to time point was used. When 4 month was not available last prior was used.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Arm I (Intervention) | Arm II (Control)
Number analyzed (Participants) | 4 | 2
cm^3 | -3.87 (8.0) | -3.045 (2.14)
Statistical Analysis 1: Comparison: Arm I (Intervention) vs Arm II (Control); Test type: Superiority or Other; p = 0.9, t-test, 2 sided

2. Primary Outcome: Change From Baseline in Peritumoral Brain Edema
Description: The relative change from baseline will be assessed longitudinally, however, the main comparison of interest is the relative change at the 4-month evaluation.For each patient change = edema at follow up - baseline edema.
Time Frame: at 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Arm I (Intervention) | Arm II (Control)
Number analyzed (Participants) | 5 | 4
cm^3 | -2.7 (7.3) | 10.21 (14.06)
Statistical Analysis 1: Comparison: Arm I (Intervention) vs Arm II (Control); Test type: Superiority or Other; p = 0.12, t-test, 2 sided

3. Primary Outcome: Change From Baseline in Peritumoral Brain Edema
Description: as for outcome 1
Time Frame: at 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Arm I (Intervention) | Arm II (Control)
Number analyzed (Participants) | 2 | 2
cm^3 | -3.7 (9.5) | -1.5 (2.9)
Statistical Analysis 1: Comparison: Arm I (Intervention) vs Arm II (Control); Test type: Superiority or Other; p = 0.8, t-test, 2 sided

4. Secondary Outcome: Quality of Life at 6 Months
Description: Quality of life as assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 Items (EORTC QLQ-C30)
Time Frame: At 2, 4, 6, 12, and 24 months
Population: At baseline and the most recent post treatment point in time, the QOL data for group 1 consist of n=3 patients and for group 2, n=2. Because of low patient numbers, no analysis was done.
Arm/Group | Arm I (Intervention) | Arm II (Control)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time-to-tumor-progression: Percentage of Patients With Tumor Progression at 6 Months
Description: Percentage of participants with tumor progression (>25% increase in tumor volume compared to time 0) will be measured from enrollment to documented progression or death whichever comes first. The method used to calculate the time to tumor progression was Kaplan Meier test method to define the 95% confidence levels.
Time Frame: 6 months
Population: All 12 patients followed to progression or death, or censored at last visit when known alive
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Intervention) | Arm II (Control)
Number analyzed (Participants) | 7 | 5
percentage of participants | 43 [-13 to 99] | 100 [100 to 100]

6. Secondary Outcome: Time-to-tumor-progression: Percentage of Patients With Tumor Progression at 1 Year
Description: as for outcome 5
Time Frame: 1 year
Population: All 12 patients followed to progression or death, or censored at last visit when known alive
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Intervention) | Arm II (Control)
Number analyzed (Participants) | 7 | 5
percentage of participants | 71 [32 to 111] | 80 [41 to 119]

7. Secondary Outcome: Overall Survival: Percentage of Patients That Were Alive at 1 Year
Description: Overall survival will be measured from the date of enrollment to date of death or last contact. Survival will be evaluated by the Kaplan Meier method to evaluate the median survival and 1 year survival rates.
Time Frame: 1 year.
Population: All 12 patients followed to death or censored at last visit when known alive
Measure: Number (95% Confidence Interval); unit: percentage of particpants
Arm/Group | Arm I (Intervention) | Arm II (Control)
Number analyzed (Participants) | 7 | 5
percentage of particpants | 57 [9 to 106] | 60 [5 to 115]

8. Other Pre Specified Outcome: Food Intake as Assessed by the Block 98 Food Frequency Questionnaire and a 3-day Food Record
Description: The 3-day food diary will be used to assess the dietary intake and to increase eating awareness of patients.
Time Frame: At 2, 4, 6, 12, and 24 months
Population: No data collected
Arm/Group | Arm I (Intervention) | Arm II (Control)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a 4 year period while patients were on treatment
Arm/Group | Arm I (Intervention) | Arm II (Control)
Serious Adverse Events (participants affected / at risk) | 0/7 | 2/5
Other Adverse Events (participants affected / at risk) | 3/7 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Intervention) (N=7) | Arm II (Control) (N=5)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) — Unrelated to intervention
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1) — Unrelated to intervention
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Intervention) (N=7) | Arm II (Control) (N=5)
Tiredness (General disorders) | 2 | 2
Heartburn (Gastrointestinal disorders) | 1 | 0
Skin Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Weight Loss (General disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0
Radiation Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1
Shingles (Skin and subcutaneous tissue disorders) | 1 | 0
Cushingoid appearance (Endocrine disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Thrush (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Rectal bleeding (Gastrointestinal disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0
Ataxia (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Mood alteration-anxiety, agitation (Psychiatric disorders) | 2 | 1
Neuropathy-sensory (Nervous system disorders) | 1 | 0
Disoriented; cries easily; angry (Psychiatric disorders) | 1 | 0
Neck pain (Nervous system disorders) | 0 | 1
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Certain outcome analysis not done due to low patient accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes